CLINICAL TRIAL: NCT02466165
Title: Multiple Sclerosis: Associated Cardiometabolic Risks and Impact of Exercise Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bert Op't Eijnde (Other)
Responsible Party: Sponsor-Investigator, Bert Op't Eijnde, PhD, Hasselt University
Organization: Hasselt University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-CMR
Record Dates: First submitted 2015-03-09; First posted 2015-06-09 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Multiple Sclerosis; Healthy Controls
Keywords: cardiometabolic risk; physical exercise
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MS patients intervention group (Experimental): the feasibilty and influence of high intense interval exercise on the cardiometabolic risk state in MS patients will be investigated in a pilot trial.
  Interventions: Behavioral: Physical exercise
- healthy controls (No Intervention): To identify whether MS patients have a higher cardiometabolic risk state than healthy controls, this project discovers the prevalence of cardiometabolic risk factors (dyslipidemia, hypertension, body fat, glucose tolerance/IR, inflammation and heart function), in MS and referent subjects.
- larger group of MS patients (No Intervention): To identify whether MS patients have a higher cardiometabolic risk state than healthy controls, this project discovers the prevalence of cardiometabolic risk factors (dyslipidemia, hypertension, body fat, glucose tolerance/IR, inflammation and heart function), in MS and referent subjects.

INTERVENTIONS:
Behavioral: Physical exercise
  Other Names: combined (endurance and resistance) exercise programme
  Arms: MS patients intervention group

SUMMARY:
Multiple Sclerosis (MS) is the most common chronic inflammatory neurological disorder in young adults. Due to heterogeneous symptoms, MS patients are often more inactive than healthy controls, resulting in an inactivity related physiological profile. In healthy people, physical inactivity can contribute to the development of an increased cardiometabolic risk state including the combined presence of cardiovascular risk factors (increased cholesterol, elevated blood pressure, body fat, glucose intolerance/insulin resistance, inflammation and reduced heart function/autonomic control). In other populations, these secondary health complications can be, in part, reduced by physical exercise, which is often used as the primary treatment strategy. Since the impact of exercise on cardiovascular risk factors in MS is unknown the present project first aims to explore this in a pilot trial and a controlled research setting (during 12 weeks). A better understanding of the above described risk factors and underlying physiological mechanisms will reduce the incidence of preventable comorbidities in MS and will further improve the multidisciplinary treatment of MS patients and MS rehabilitation in particular. Interestingly, the investigators already reported an elevated prevalence of impaired glucose tolerance in MS, but it is not clear whether the cardiometabolic state in MS is also impaired. Therefore, in a second part, the researchers will explore whether MS patients present a higher risk to develop cardiovascular diseases, as measured by the assessment of various cardiovascular risk factors, compared to healthy controls.

DETAILED DESCRIPTION:
In a first part, various cardiovascular risk factors will be determined in a group of MS patients (n=~16). These patients will be enrolled in a pilot trail, investigating the feasability and impact of a high intense interval exercise intervention (12 weeks high intensity interval training). After 12 weeks, baseline cardiovascular risk measurements will be repeated to determine the impact of high intensity interval training on these risk factors in MS.

In a second part, these cardiovascular risk factors in a larger group of MS patients (n=~50) will be compared to healthy controls (n=~25), in order to determine whether MS patients show an increased prevalence of cardiovascular risk factors, and thus an elevated risk to develop cardiovascular diseases.

In total, a group of 80 subjects (MS patients and HC) will be investigated throughout this study, with only MS patients participating in the pilot trial/exercise intervention.

Measurements of cardiovascular risk factors will include:

* body composition (DEXA)
* blood pressure and heart rate (Omron M4-I)
* whole body glucose disposal (oral glucose tolerance test)
* blood analysis: insulin, total cholesterol, high- density lipoprotein, low-density lipoprotein, plasma triglycerides, C-reactive protein and glycosylated haemoglobin.

Furthermore, a maximal exercise test (determination maximal heart rate, workload, lactate concentrations, etc) and an isometric/isokinetic strength test will be performed to determine the impact of the rehabilitation program in MS patients.

ELIGIBILITY:
Inclusion Criteria:

Healthy controls:

* male/female
* 18 years
* written informed consent (Declaration of Helsinki and ethical committee guidelines)

MS patients:

* cfr healthy controls criteria, in addition:
* Diagnosed MS according to the McDonald criteria
* Expanded Disability Status Scale (EDSS) between 1 and 7
* Being available for the complete study course

Exclusion Criteria:

* other disorders
* pregnancy
* participation in another study
* MS exacerbation 6 months prior to the start.
* for the MS patients: contra-indication to perform physical exercise

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
dyslipidemia, as determined by the analysis of blood samples | change from baseline up to 12 weeks
  measured at baseline and after 12 of exercise Blood samples will be analysed to determine complete blood lipid profile.
hypertension / blood pressure as determined by supine blood pressure measures | change from baseline up to 12 weeks
  measured at baseline and after 12 of exercise Blood pressure will be evaluated supine.
body fat as determined by DEXA scan | change from baseline up to 12 weeks
  measured at baseline and after 12 weeks of exercise Body composition will be determined by means of a Dexa scan.
glucose tolerance / insulin resistance as determined by oral glucose tolerance test | change from baseline up to 12 weeks
  measured at baseline and after 12 weeks of exercise Glucose tolerance will be evaluated by means of an oral glucose tolerance test. Collected blood samples will be analysed to determine insulin concentrations
inflammation as determined by analysis of blood samples | change from baseline up to 12 weeks
  measured at baseline and after 12 weeks of exercise Blood samples, as collected during the oral glucose tolerance test, will be analysed to evaluate inflammation (CRP etc)

SECONDARY OUTCOMES:
muscle strength of knee extensor/flexor and elbow extensor/flexor as determined by Biodex | change from baseline up to 12 weeks
  measured at baseline and after 12 weeks of exercise Muscle strength will be evaluated by means of the Biodex
aerobic capacity as determined by a maximal endurance test on the bike | change from baseline up to 12 weeks
  measured at baseline and after 12 weeks of exercise Aerobic capacity will be tested during a maximal endurance test on the bike
blood lactate concentrations during exercise as determined by a maximal endurance test on the bike | change from baseline up to 12 weeks
  measured at baseline and after 12 weeks of exercise Lactate concentrations (mmol/L) will be tested during a maximal endurance test on the bike
heart function | change from baseline up to 12 weeks
  measured at baseline and after 12 and 24 weeks of exercise

CONTACTS AND LOCATIONS:
Overall Officials: Bert O Eijnde, Ph.D., Study Chair — Hasselt University, REVAL/BIOMED
Locations (2):
- Belgium (2):
  - REVAL, Diepenbeek
  - Jessa hospital, Hasselt